CLINICAL TRIAL: NCT00885092
Title: Wettability of Silicone Hydrogel Lenses With SiH MPDS FID 114675A vs. A Marketed Multi-Purpose Solution
Brief Title: Single Site Study of the Wettability of Contact Lenses With an Investigational Multi-Purpose Disinfecting Solution vs. a Marketed Multi-Purpose Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: C-08-082
Record Dates: First submitted 2009-04-17; First posted 2009-04-21 (Estimated); Results first posted 2012-03-20 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Contact Lens Care
Keywords: Contact lenses; Disinfecting solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 114675A / RepleniSH (Other): FID 114675A in Period 1; RepleniSH in Period 2. Each solution was used for 7 days for cleaning, rinsing, conditioning, disinfecting, and storing silicone hydrogel contact lenses, per protocol-specified instructions. A new pair of silicone hydrogel contact lenses was dispensed at the start of each period and worn bilaterally on a daily wear basis.
  Interventions: Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS); Device: RepleniSH Multi-Purpose Disinfecting Solution (MPDS) (OPTI-FREE® RepleniSH®); Device: Senofilcon A contact lens (ACUVUE® Oasys™); Device: Balafilcon A contact lens (PureVision®)
- RepleniSH / FID 114675A (Other): RepleniSH in Period 1; FID 114675A in Period 2. Each solution was used for 7 days for cleaning, rinsing, conditioning, disinfecting, and storing silicone hydrogel contact lenses, per protocol-specified instructions. A new pair of silicone hydrogel contact lenses was dispensed at the start of each period and worn bilaterally on a daily wear basis.
  Interventions: Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS); Device: RepleniSH Multi-Purpose Disinfecting Solution (MPDS) (OPTI-FREE® RepleniSH®); Device: Senofilcon A contact lens (ACUVUE® Oasys™); Device: Balafilcon A contact lens (PureVision®)

INTERVENTIONS:
Device: FID 114675A Multi-Purpose Disinfecting Solution (MPDS) — Investigational solution intended for use as a cleaning, rinsing, conditioning, disinfecting, and storage solution for silicone hydrogel (SiH) contact lenses.
Device: RepleniSH Multi-Purpose Disinfecting Solution (MPDS) (OPTI-FREE® RepleniSH®) — Commercially marketed solution intended for use as a cleaning, conditioning, rinsing, disinfecting, and storage solution for all silicone hydrogel and soft (hydrophilic) contact lenses.
  Other Names: (OPTI-FREE® RepleniSH®)
Device: Senofilcon A contact lens (ACUVUE® Oasys™) — Commercially marketed silicone hydrogel contact lens for daily wear use
  Other Names: ACUVUE® Oasys™
Device: Balafilcon A contact lens (PureVision®) — Commercially marketed silicone hydrogel contact lens for daily wear use
  Other Names: PureVision®

SUMMARY:
The purpose of this study is to clinically evaluate an investigational multi-purpose disinfecting solution (MPDS) compared to a commercial MPDS with respect to wettability of silicone hydrogel contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Must be successfully wearing assigned study lens brand (either ACUVUE® OASYS™ or PureVision® contact lenses) for at least 7-10 days, minimum 8 hours a day, prior to Visit 1 (screening).
* Vision correctable to 20/30 (Snellen) or better in each eye at distance with study lenses at Visit 1 (screening).
* Must have discontinued contact lens wear for at least two consecutive days before Visit 2 (baseline).
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any medical condition (systemic or ophthalmic) that may, in the opinion of the investigator, preclude safe administration of test article or safe participation in the study.
* Known sensitivity or intolerance to any protocol-specified contact lens solutions, eye drops, or products containing similar ingredients (e.g., generic products).
* Monocular vision (only one eye with functional vision) or fit with only one contact lens.
* Use of topical ocular over-the-counter or prescribed topical ocular medication, with the exception of rewetting drops, within 7 days prior to screening visit.
* Current or history of ocular infection, inflammation, disease, structural abnormality or conditions within the last 6 months that could affect study participation or may preclude safe administration of the investigational lens care solution, in the opinion of the investigator.
* Any corneal surgery, cataract surgery, intraocular lens implants or glaucoma filtering surgery within the last 12 months.
* Any slit-lamp finding score of 1 (or rated 3 or 4 for limbal and bulbar conjunctival injection) at screening or baseline visits.
* Corneal staining area assessment ≥ 20% in any corneal region in either eye at screening or baseline visit.
* Corneal staining graded as 2 (macropunctate) or greater in any corneal region in either eye at baseline visit.
* Participation in any investigational clinical study within 30 days of baseline visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one US study center.
Pre-assignment Details: 40 participants with normal eyes (other than vision correction) were enrolled in the trial. After the screening visit, participants discontinued contact lens wear and wore their glasses for at least 2 days as a washout prior to Period 1. A similar washout occurred prior to Period 2. Cross-over study design.
Groups:
- FID 114675A / RepleniSH: FID 114675A in Period 1; RepleniSH in Period 2. Each solution was used for 7 days, per protocol-specified instructions. A new pair of silicone hydrogel contact lenses was dispensed at the start of each period and worn bilaterally on a daily wear basis.
- RepleniSH / FID 114675A: RepleniSH in Period 1; FID 114675A in Period 2. Each solution was used for 7 days, per protocol-specified instructions. A new pair of silicone hydrogel contact lenses was dispensed at the start of each period and worn bilaterally on a daily wear basis.
Period: Period 1, 7 Days
Arm/Group | FID 114675A / RepleniSH | RepleniSH / FID 114675A
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Period 2, 7 Days
Arm/Group | FID 114675A / RepleniSH | RepleniSH / FID 114675A
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FID 114675A / RepleniSH: FID 114675A in Period 1; RepleniSH in Period 2. Each solution was used for 7 days, per protocol-specified instructions. Contact lenses worn bilaterally on a daily wear basis, with a new pair dispensed at the beginning of each period.
- RepleniSH / FID 114675A: RepleniSH in Period 1; FID 114675A in Period 2. Each solution was used for 7 days, per protocol-specified instructions. Contact lenses worn bilaterally on a daily wear basis, with a new pair dispensed at the beginning of each period.
- Total: Total of all reporting groups
Arm/Group | FID 114675A / RepleniSH | RepleniSH / FID 114675A | Total
Number analyzed (Participants) | 20 | 20 | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.1) | 42.4 (10.0) | 42.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Ex-Vivo Wetting Angle
Description: Study lens was removed from the eye according to protocol-specified procedures. The OCA15 (Optical Contact Angle) Instrument was used to observe, record, and calculate contact angle measurements. The wetting angle measurement was recorded in degrees (0-180), and a lower wetting angle measurement indicates a more wettable lens.
Time Frame: Day 7, Hour 14
Population: Intent to treat: All participants who received regimen and had at least one on-therapy visit. Cross-over study design.
Measure: Mean (Standard Deviation); unit: Degrees
Groups:
- FID 114675A: FID 114675A solution used 7 days for cleaning, rinsing, conditioning, disinfecting, and storing silicone hydrogel contact lenses, per protocol-specified instructions. A new pair of silicone hydrogel contact lenses was dispensed at the start of the 7 days and worn bilaterally on a daily wear basis.
- RepleniSH: Commercially marketed solution used 7 days for cleaning, rinsing, conditioning, disinfecting, and storing silicone hydrogel contact lenses, per protocol-specified instructions. A new pair of silicone hydrogel contact lenses was dispensed at the start of the 7 days and worn bilaterally on a daily wear basis.
Arm/Group | FID 114675A | RepleniSH
Number analyzed (Participants) | 40 | 40
Degrees | 52.1 (32.7) | 59.6 (38.1)

2. Secondary Outcome: Mean Lens Comfort
Description: Lens comfort was assessed by the participant on a 5-point Likert scale prior to any examination. The participant was instructed to select a single response to the statement, "My lenses feel comfortable right now," with 1 = strongly disagree, 2 = disagree, 3 = undecided, 4 = agree, and 5 = strongly agree.
Time Frame: Day 7, Hour 14
Population: Intent to treat: All participants who received regimen and had at least one on-therapy visit. Cross-over study design.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FID 114675A | RepleniSH
Number analyzed (Participants) | 40 | 40
Units on a scale | 4.1 (0.9) | 3.8 (0.9)

3. Secondary Outcome: Percentage of Participants With Solution-Related Corneal Staining
Description: Corneal staining was assessed by the investigator using fluorescein dye, a yellow filter, and a slit lamp. Corneal staining was graded on a continuous scale of 0% (no staining in the region) to 100% (staining covers entire region) in 1% increments for 5 corneal regions (central, nasal, temporal, inferior, and superior). Solution-related corneal staining was defined as ≥20% corneal staining area in at least 3 corneal regions of both eyes and is reported as a percentage of total participants.
Time Frame: Day 7, Hour 14
Population: Intent to treat: All participants who received regimen and had at least one on-therapy visit. Cross-over study design.
Measure: Number; unit: Percentage of participants
Arm/Group | FID 114675A | RepleniSH
Number analyzed (Participants) | 40 | 40
Percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 24 March 2009 to 5 May 2009.
Description: This reporting group includes all participants enrolled and exposed to test regimen.
Groups:
- FID 114675A: FID 114675A solution used 7 days for cleaning, rinsing, conditioning, disinfecting, and storing silicone hydrogel contact lenses, per protocol-specified instructions.
- RepleniSH: Commercially marketed solution used 7 days for cleaning, rinsing, conditioning, disinfecting, and storing silicone hydrogel contact lenses, per protocol-specified instructions.
Arm/Group | FID 114675A | RepleniSH
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes